CLINICAL TRIAL: NCT03623685
Title: RANDOMİZED , PROSPEKTİVE COHORT STUDY FOR UTEROCERVİCAL ANGLE MEASUREMENT BY ULTRASOUND FOR PREDİCTİNG SPONTANEOUS PRETERM BİRTH
Brief Title: UTEROCERVİCAL ANGLE MEASUREMENT IN SPONTANEOUS PRETERM BIRTH (UAMSPB)
Acronym: UAMSPB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Istanbul Medeniyet University (Other)
Collaborators: Meryem Dilara Yetimoğlu (Unknown); İdris Yetimoğlu (Unknown)
Responsible Party: Principal Investigator, Özkan Özdamar, associate professor, Istanbul Medeniyet University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2017/0343
Record Dates: First submitted 2018-07-24; First posted 2018-08-09 (Actual); Last update posted 2018-08-09 (Actual); Status verified 2018-08

CONDITIONS: Preterm Labor
Keywords: uterocervical angle; preterm labor
MeSH Terms: conditions — Obstetric Labor, Premature

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- voluson 8 (Experimental)
  Interventions: Diagnostic Test: measurement of uterocervical angle

INTERVENTIONS:
Diagnostic Test: measurement of uterocervical angle — We will measure between internal cervikal os and external cervical os. After we will draw a line between anterior uterine wall and internal cervical os. Then we will measure angle between two lines

SUMMARY:
İn this study Study; Between August 2018 and August 2019, the Ministry of Health, Medeniyet University, Göztepe Training and Research Hospital, Gynecology and Obstetrics Clinic Will be Included for Routine Control Purposes, Single Pregnancies Between 16-24 Weeks and no Known Risk Factors for Preterm Delivery . Each Participant Will be Given Written and Verbal Information About the Work and Will be Informed. Uterocervical Angle Measurement; Dorsolithotomy, Using a Sterilized Vaginal Ultrasonic Probe. It Will be Seen That the Distance Between the Internal Cervical os and the External Cervical os is Inclusive of the Cervical Isthmus That Can be Seen With the Anterior Uterine Wall. The First Line Will be Drawn Between the Internal Cervical os and the External Cervical os. The Second Line Will be Drawn as Passing Through the Internal Cervical Ostia, Parallel to the Anterior Uterine Wall. The Angle Between the Two Lines on the Internal Cervical Vertebra Will be Measured. Patients Will be Followed up Until the End of the 37th Gestational Week. The Gestation Week They Are Giving Birth Will be Recorded. Patients Were Then Classified as Before and After 37 Gestational Weeks and Uterocervical Angle Measurements Between 16-24 Gestational Weeks Were Compared.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who did not have complaints between December 2017 and August 2018, who went to polyclinic because of routine control
2. Patients who had a pregnancy between 16-24 weeks
3. Patients with singleton pregnancy
4. Patients with a cervical length of 25 mm or more

Exclusion Criteria:

1. Patients with preterm labor history (under 37 weeks) in previous pregnancy
2. Patients with premature rupture of membranes in current pregnancy
3. Patients with past uterine cervical surgery (conization, LEEP) as a cause of premature birth
4. Patients with preterm birth
5. Placenta anomalies present pregnancy
6. Patient with retrovert uterus, uterine fibroid of lower segment

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2 (Estimated)
Dates: Start 2018-08-10 (Estimated); Primary Completion 2019-08-10 (Estimated); Study Completion 2019-12-10 (Estimated)

PRIMARY OUTCOMES:
The measurement of patients after they give birth | 1 year
  Images were re-measured for uterocervical angle between the lower uterine segment and the cervical canal. Primary outcome was prediction of <37 weeks by uterocervikal angle.

CONTACTS AND LOCATIONS:
Overall Officials: özkan özdamar, Principal Investigator — Istanbul Medeniyet University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dziadosz M, Bennett TA, Dolin C, West Honart A, Pham A, Lee SS, Pivo S, Roman AS. Uterocervical angle: a novel ultrasound screening tool to predict spontaneous preterm birth. Am J Obstet Gynecol. 2016 Sep;215(3):376.e1-7. doi: 10.1016/j.ajog.2016.03.033. Epub 2016 Mar 24. PMID 27018466